CLINICAL TRIAL: NCT06240091
Title: An Exploratory Open-Label Potency and Precision Investigation of a Relational Agent Intervention
Brief Title: Potency and Precision Investigation
Acronym: PAPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woebot Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: W-DISC-002
Record Dates: First submitted 2024-01-23; First posted 2024-02-02 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Depression, Anxiety
Keywords: Woebot; Relational agent; Digital mental health intervention; Chatbot; Conversational agent; Natural language processing; Artificial intelligence
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- DISC-MA (Experimental): All participants will be asked to download and use the DISC-MA study application. They will have access to the app throughout the 4 week study.
  Interventions: Device: DISC-MA

INTERVENTIONS:
Device: DISC-MA — DISC-MA is a digital program that utilizes elements from validated psychotherapies (e.g., cognitive behavioral therapy), with a relational agent (Woebot) that engages users in conversations with responses that are selected from a list based on natural language processing.

SUMMARY:
The overarching goal of this study is to establish initial proof of mechanism for precision interventions in an adult population.

DETAILED DESCRIPTION:
This exploratory single-arm trial will provide initial learning on the current implementation of precision interventions and generate data and hypotheses to inform the exploration of future interventions by identifying mechanisms and moments in the user journey to target. The DISC-MA app uses a relational agent (Woebot) to engage users in conversations. Eligible participants will be assigned to use DISC-MA, in which Woebot selects from a list of responses based on natural language processing. Participants will receive instructions on downloading and using the DISC-MA app in order to access the intervention. Participants will use the app as instructed and will complete assessments for the primary endpoint as Week 4 (EOT) with additional measures being collected as Baseline, Week 1, and Week 2. Results from this study will provide data on baseline participant clinical and psychological characteristics and their engagement with DISC-MA, and associations between the two.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18-75 years of age
2. Must own or have regular access to a smartphone with a recent operating system installed (Android: OS 8.0 or higher, Apple: iOS 13.0 or higher) with reliable Wi-Fi access or sufficient data plan to engage with assigned treatment condition for the duration of the study
3. Must be available and committed to engage with the program and complete assessments for a 4-week duration
4. Must be able to read and write in English
5. Must have primary residence in the United States
6. Must have mild or greater symptoms of depression and/or anxiety at Screening/Baseline, indicated by a score > 4 on the Patient Health Questionnaire (PHQ-8) and/or Generalized Anxiety Disorder (GAD-7)

Exclusion Criteria:

1. Current suicidal ideation with a plan and/or intent or a suicide attempt within the past 12 months
2. Previous Woebot use
3. Involuntary inpatient psychiatric hospitalization any time within the past 30 days
4. Lifetime diagnosis of bipolar disorder
5. Lifetime diagnosis of a psychotic disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Campellone, PhD, Principal Investigator — Woebot Health
Locations (1):
- Woebot Investigational Site, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DISC-MA
Started | 203
Completed | 201
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | DISC-MA
Number analyzed (Participants) | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.22 (13.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154
  Male | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latinx | 21
  Non-Hispanic American Indian or Alaskan Native | 1
  Non-Hispanic Asian | 16
  Non-Hispanic Black or African American | 38
  Non-Hispanic Middle Eastern or North African | 2
  Non-Hispanic more than one race | 11
  Non-Hispanic White | 114
Region of Enrollment [Number; unit: participants]
  United States | 203

OUTCOME MEASURES:

1. Primary Outcome: Working Alliance Inventory-Short Revised (WAI-SR), Total Scale
Description: Measure of working alliance. A 12-item measure that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy, and (c) development of an affective bond. For the purposes of the study, the word "therapist" was replaced with "Woebot". Total mean scores range from 1-5, with higher scores indicating greater alliance between the participant and Woebot.
Time Frame: 1 week and Post-treatment at 4 weeks
Population: Data missing
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DISC-MA
Number analyzed (Participants) | 201
score on a scale
  Week 1 Goal: number analyzed (Participants) | 192
  Week 1 Goal | 3.63 (0.98)
  Week 1 Task: number analyzed (Participants) | 192
  Week 1 Task | 3.25 (0.88)
  Week 1 Bond: number analyzed (Participants) | 192
  Week 1 Bond | 3.95 (0.96)
  Week 1 Total: number analyzed (Participants) | 192
  Week 1 Total | 3.61 (0.83)
  Week 4 Goal: number analyzed (Participants) | 188
  Week 4 Goal | 3.72 (0.99)
  Week 4 Task: number analyzed (Participants) | 188
  Week 4 Task | 3.40 (0.92)
  Week 4 Bond: number analyzed (Participants) | 188
  Week 4 Bond | 4.02 (0.98)
  Week 4 Total: number analyzed (Participants) | 188
  Week 4 Total | 3.71 (0.87)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | DISC-MA
All-Cause Mortality (participants affected / at risk) | 0/203
Serious Adverse Events (participants affected / at risk) | 2/203
Other Adverse Events (participants affected / at risk) | 56/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DISC-MA (N=203)
Eating disorders and disturbances (Psychiatric disorders) | 1 (1)
Active suicidal ideation (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DISC-MA (N=203)
Psychiatric disorders (Psychiatric disorders) | 25 (37)
General disorders (General disorders) | 4 (4)
Surgical and medical procedures (Surgical and medical procedures) | 1 (1)
Prostatic disorder (Reproductive system and breast disorders) | 2 (2)
Nervous system disorders (Nervous system disorders) | 4 (4)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 6 (6)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 3 (4)
Investigations (Investigations) | 2 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2)
Glaucoma (Eye disorders) | 1 (1)
Chiari malformation (Congenital, familial and genetic disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Pre-diabetic (Metabolism and nutrition disorders) | 1 (1)
Parathyroid tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Surgical wound (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT06240091/Prot_SAP_000.pdf